CLINICAL TRIAL: NCT05621122
Title: Characterizacion of Pro-VEgetarian Diets: Diet Quality and Nutrition, MIcrobial/Metabolite Profiles and Implications in CAncer (MIVECA Study)
Brief Title: Pro-Vegetarian Diets, Microbial/Metabolite Profiles and Cancer
Acronym: MIVECA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Andalusian School of Public Health (Other Government); Institut Investigacio Sanitaria Pere Virgili (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); National Research Council, Spain (Other Government); Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government); University of Seville (Other); Biodonostia Health Research Institute (Biodonostia HRI) (Unknown)
Responsible Party: Principal Investigator, Esther Molina-Montes, Professor (Assistant), Universidad de Granada
Other Study IDs: PPJIA2021-38
Record Dates: First submitted 2022-09-29; First posted 2022-11-17 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Dietary Habits; Food Habits; Nutrition, Healthy; Cancer; Metabolic Disease
Keywords: dietary patterns; vegetarian; omics; microbiome; cancer; metabolism
MeSH Terms: conditions — Feeding Behavior; Neoplasms; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Omnivours: 100 subjects (comparison group)
  Interventions: Other: This is an observational study
- Vegans: 50 subjects, adults aged over 18 years, voluntarly participating in this observational study
  Interventions: Other: This is an observational study
- Lacto-ovo-vegetarians: 50 subjects, adults aged over 18 years, voluntarly participating in this observational study
  Interventions: Other: This is an observational study
- Pesco-vegetarians: 50 subjects, adults aged over 18 years, voluntarly participating in this observational study
  Interventions: Other: This is an observational study
- Pro-vegetarians: 50 subjects, adults aged over 18 years, voluntarly participating in this observational study
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study. The control group (omnivours) will be compared with all otgher groups

SUMMARY:
This projects aims to characterize dietary habits and nutrition quality of pro-vegetarian diets as compared to omnivorous diets. It also aims to stablish gut microbial and metabolit profiles of this dietary pattern, in order to elucidate the role of plant-based diets in cancer prevention and treatment.

DETAILED DESCRIPTION:
Plant-based foods (fruits, vegetables, cereals, nuts and seeds, legumes, and vegetable oils) are the main source of fiber and other bioactive compounds in the diet. Plant-based diets are therefore assumed to prevent mortality and the ocurrence of chronic diseases including cancer. However, evidence on this issue is still scarce, and the mechanisms and drivers of their potential health benefits are also only partially known.

The main objectices of this project are:

1. To develop and validate dietary assessment methods for the vegetarian population
2. To assess dietary habits and consumer beliefs of vegetarians with respect to omnivores, considering different types of vegetarian diets
3. To identify a gut microbiota signature related to plant-based diets from subgroups of subjects following a plant-based diet foods (vegans, lacto-vegetarians, …, and pro-vegetarians) and omnivorous subjects (non-plant-based diets), from stool metagenomic sequencing.
4. To relate this signature with metabolites present in faeces (related to the presence of certain microbial species) and in urine to improve the predictive capacity of the microbial signature of vegetable diets.
5. Validate the signature using independent study populations, and including colorectal and breast cancer survivors as another study target.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* pregnancy or lactation
* antibiotic treatment in the previous 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University students and staff, mainly. Healthy volunteers from the general population. The control group will be matched by age and sex to the vegetarian diet study groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary habits obtention from vegetarians: the dietary intake | 3 months
  Dietary habits will be taken by an online specific Food Frequency Questionnaire (FFQ) for Spanish population, including novel vegetarian foods to evaluate vegetarian food consumption. The data analysis will be taken at baseline outcome.
Dietary assessment validation methods: 24-hour-recalls and dietary intake biomarkers | 6 monts
  To validated dietary assessment method, two 24-Hour-Recalls in two non-consecutive days will be used, as well as the analysis of specific vegetarian diet metabolites in urine and stool samples using Ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS). The data analysis will be taken at baseline. We have estimated that 200 subjects will be sufficient to detect, with a 95% confidence and power of 90%, correlation coefficients greater than rho=0.2.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Molina Montes, Study Director — Universidad de Granada; Noelia M Rodriguez, Study Chair — nmrodriguez@ig.csic.es
Locations (6):
- Spain (6):
  - Idibell Ico, Barcelona
  - Biodonostia, Donostia / San Sebastian
  - University of Granada, Granada
  - Csic-Ictan, Madrid
  - CSIC-IG, Seville
  - IISPV Pere Virgili, Tarragona

IPD SHARING:
Plan to Share IPD: No